CLINICAL TRIAL: NCT05855707
Title: Wharton's Jelly Mesenchymal Stromal Cell (WG-MSC) Injections as GVHD Prophylaxis in Hematopoietic Allogeneic Stem Cell Transplantation With an Haplo-identical Donor : a Dose Escalation Study
Brief Title: Wharton Jelly Mesenchymal Stromal Cells as GVHD Prophylaxis
Acronym: HAPLO-GEL
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Saint-Louis Hospital, Paris, France (Other)
Responsible Party: Principal Investigator, Maud D'AVENI, MCU-PH, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2023-504268-40-00
Record Dates: First submitted 2023-05-04; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Allogeneic Disease; GVHD,Acute; Graft Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- maximum tolerated dose (Experimental): 1. x10e6 WJ-MSC/kg/infusion for 3 weekly infusions 1.5x10e6 WJ-MSC/kg/infusion for 3 weekly infusions
  2. x10e6 WJ-MSC/kg/infusion for 3 weekly infusions
  Interventions: Biological: WJ-MSC infusion

INTERVENTIONS:
Biological: WJ-MSC infusion — cellular therapy

SUMMARY:
Despite progress in chemotherapy, targeted therapy and immunotherapy, allogeneic hematopoietic stem cell transplantation (allo-SCT) is still the only curative procedure for some hematological malignancies. The probability of finding a matched sibling donor (MSD) is estimated under the classical 30%, because of the age of patients and their relatives, and a matched unrelated donor (MUD) can take time to identify. Currently in France, 25% of the allo-SCT are performed with an haplo-identical related donor. The Baltimore group developed an approach using haploidentical related donors, RIC, T-replete bone marrow and post-transplant high dose cyclophosphamide (PTCy) in patients with advanced hematological malignancies. PTCy has shown to eradicate alloreactive donor and host T-cells, activated by respective antigens, thereby reducing the incidence of graft versus host disease (GvHD) but delaying hematopoietic recovery. Therefore, the main source of graft is peripheral blood stem cells (PBSC) mobilized by G-CSF in France. Unfortunately, with PBSC we observe a higher cumulative incidence of GvHD (around 50%) and a higher toxicity-related mortality (TRM), especially for recipients >50 years old. The co-transplantation of Mesenchymal Stem Cells (MSC) at the time of transplantation has previously shown a double interest in GvHD immunomodulation and hematopoiesis support. Pre-clinical studies (in mice) have shown that mesenchymal stromal cells (MSCs) from Wharton's Jelly reduce the incidence of GvHD when the infusions are weekly repeated. We propose a phase I clinical trial to find the maximum tolerated dose (MTD) of a weekly infusion of WJ-MSC administered as GvHD prophylaxis and as a support for a faster hematological reconstitution after haplo-identical allo-SCT.

ELIGIBILITY:
Inclusion Criteria:

* With AML/ALL/SMD/SMP or lymphoid neoplasm requiring allogeneic stem cell transplantation
* In complete response (CR) for AML/ALL or CR,partial response (PR) or non pre-treated for SMD/SMP and lymphoid neoplasm
* Without a HLA matched related donor available and with identification of a haploidentical donor (brother, sister, parents, adult children or cousin)

With usual criteria for HSCT:

* ECOG ≤ 2
* No severe and uncontrolled infection
* Cardiac function compatible with high dose of cyclophosphamide
* Adequate organ function: ASAT and ALAT ≤ 2N, total bilirubin ≤ 1.5N, creatinine clearance ≥30ml/min (except if those abnormalities are linked to the hematological disease)

  * Requiring a RIC or non myeloablative conditioning:

    (i) >50 years old; (ii) heavily pre-treated; (iii) Comoribidities according to Sorror et al. Blood 2005;106(8):2912-9, notamment HCT/CI≥ 3 (JAMA. 2011 Nov 2;306(17):1874-83).
  * With health insurance coverage (bénéficiaire ou ayant droit)
  * Understand informed consent or optimal treatment and follow-up
  * Contraception methods must be prescribed during all the duration of the research and using effective contraceptive methods during treatment and within 12 months for women of childbearing age and 6 months for men of childbearing age after the last dose of cyclophosphamide

Exclusion Criteria:

* History of Cancer in the last 5 years
* Uncontrolled infection: Seropositivity for HIV or HTLV-1 or active hepatitis B or C defined by a positive PCR HBV or HCV and hepatic cytolysis due to HBV
* Uncontrolled coronary insufficiency, recent myocardial infarction <6 month, current manifestations of heart failure, uncontrolled cardiac rhythm disorders, ventricular ejection fraction <50%
* Pulmonary failure with DLCO<50%
* Addition of immunosuppressant treatment for GVHD prophylaxis (except immunosuppressant allowed per protocol)
* Renal failure with creatinine clearance <50ml / min
* Pregnancy (β-HCG positive) or breast-feeding
* Any debilitating medical or psychiatric illness which would preclude the realization of the SCT or the understanding of the protocol
* Under protection by law (tutorship or curatorship)
* Unwilling or unable to comply with the protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 7 days
  The maximum tolerated dose (MTD) will be defined by the highest dose (highest level) where no patient out of 3, or only 1 patient out of 6 presents with dose-limiting toxicity (DLT).
  The occurrence, within 7 days following one of the three injections, of any adverse event (AE) reasonably related to the injection of CSM-GW grade 3 to 5 according to the NCI-CTCAE classification version 5.0, or part of the "Important Medical Event list", or having a severity criterion
  The maximum tolerated dose (MTD) will be defined by the highest dose (highest level) where no patient out of 3, or only 1 patient out of 6 presents with dose-limiting toxicity (DLT).
  The occurrence, within 7 days following one of the three injections, of any adverse event (AE) reasonably related to the injection of CSM-GW grade 3 to 5 according to the NCI-CTCAE classification version 5.0, or part of the "Important Medical Event list", or having a severity criterion

SECONDARY OUTCOMES:
acute and chronic GVHD incidence | 12 months
toxicity-related mortality (TRM) | 12 months
relapse incidence (RI) | 12 months
overall surival (OS) | 12 months
GvHD and relapse free survival (GRFS) | 12 months
poor graft function | 12 months

IPD SHARING:
Plan to Share IPD: Undecided